CLINICAL TRIAL: NCT02544724
Title: Single-Arm, Open-Label Study To Evaluate The Safety, Tolerability And Preliminary Efficacy Of NM-IL-12 (rHuIL-12) In Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL) Undergoing Salvage Chemotherapy
Brief Title: NM-IL-12 (rHuIL-12) In Relapsed/Refractory Diffuse Large B- Cell Lymphoma (DLBCL) Undergoing Salvage Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neumedicines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM-ONC-002
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse (DLBCL)
Keywords: Relapsed; Refractory; DLBCL; Chemotherapy
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NM-IL-12 (Experimental): NM-IL-12 will be administered subcutaneously
  Interventions: Biological: NM-IL-12

INTERVENTIONS:
Biological: NM-IL-12 — Single SC administration of NM-IL-12 will be administered at least 48 hours after completion of the last chemotherapy dose of each cycle
  Other Names: rHu-IL12

SUMMARY:
NM-IL-12 is being evaluated as an immunotherapeutic with concomitant hematopoietic regenerating properties for treatment of relapsed/refractory DLBCL, an aggressive type of B-cell non-Hodgkin's lymphoma (NHL). Determination of the maximum tolerated dose (MTD) for NM-IL-12 is not planned in this study, rather, a pre-defined dose of 150 ng/kg will be explored; this dose is based on two safety and tolerability studies of NM-IL-12 in healthy volunteers.

DETAILED DESCRIPTION:
This is a single-arm, open-label, non-randomized, multi-center study with NM-IL-12 dosed in combination with salvage chemotherapy regimens (R-ICE = rituximab plus ifosfamide-carboplatin-etoposide, R-DHAP = rituximab plus cytosine arabinoside-cisplatin-dexamethasone) for treatment of patients with relapsed/refractory DLBCL.

NM-IL-12 (150 ng/kg) will be administered subcutaneously. Patients will be monitored as routinely practiced; in addition, approximately 1 day after NM-IL-12 injection, patients will have a home visit by a nurse for blood sampling related to pharmacokinetic and pharmacodynamic (PK/PD) evaluation.

Twelve patients are planned to be enrolled into the study; initially 6 patients will be enrolled. The decision to continue and recruit the remaining six patients will be made by Data Safety Monitoring Board (DSMB) after review of relevant safety data, clinical laboratory evaluations, and vital signs collected up to 21 days post enrollment of the last patient in the first treated group. Common Terminology Grades for Adverse Events (CTCAE) guidelines will be used to determine dose-modifying criteria (DMC).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed/refractory diffuse large B- cell lymphoma (DLBCL) within 28 days prior to enrollment
2. PET/CT evaluation performed within 28 days prior to enrollment demonstrates measurable disease
3. Age >18 years
4. Eligible for intensive salvage chemotherapy with R-ICE, R-DHAP
5. Patient received first line of chemotherapy when DLBCL was initially diagnosed and did not receive any further chemotherapy until enrollment in this study
6. All treatment-related toxicities from prior chemotherapy resolved to grade ≤ 1or resolved to grade 2 only if deemed clinically not significant and approved by the Sponsor
7. ECOG performance status ≤ 2
8. Adequate organ function obtained within 28 days prior to enrollment:

   * Absolute neutrophil count ≥ 1,000/μL
   * Platelet count ≥ 50,000/μL
   * Total bilirubin ≤ 1.5x institutional upper limit of normal (IULN)
   * AST and ALT ≤ 2x IULN
   * Creatinine ≤ 2x IULN
   * Creatinine clearance ≥ 45 mL/min/1.73m2 for participants with creatinine levels above IULN
   * Albumin ≥ 2.5 g/dL
   * Prothrombin time (PT) and PTT 80% to 120% of institutional normal range
9. Women of childbearing potential must have a negative serum pregnancy test and must agree to use effective contraception, defined as intrauterine devices, double barrier method (condom plus spermicide or diaphragm) or abstain from sexual intercourse during the study
10. Male subjects must be willing to use an appropriate method of contraception (e.g., condoms) or abstain from sexual intercourse and inform any sexual partners that they must also use a reliable method of contraception (e.g., birth control pills) during the study
11. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
12. Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

1. Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose of the first cycle of the chemotherapy regimen. Infections controlled on concurrent antimicrobial agents are acceptable, and antimicrobial prophylaxis per institutional guidelines are acceptable. Patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24-48 hours prior to study enrollment
2. Known active hepatitis B or C infections, known human immunodeficiency virus (HIV) infection or known to be positive for HCV RNA or HBsAg (HBV surface antigen)
3. History of or active central nervous system (CNS) involvement by lymphoma
4. Prior or concomitant malignancy in the past 5 years that is currently active and likely to interfere with the patient's treatment for DLBCL or that is likely to increase the patient's morbidity or mortality
5. Concomitant illness associated with a likely survival of < 1 year
6. Any life-threatening illness, medical condition or organ system dysfunction that, in the investigator's opinion, could compromise the patient's safety, or put the study outcomes at undue risk
7. Prior chemotherapy or radiation therapy (unless related to NHL / DLBCL treatment) within the last 5 years
8. Cytotoxic drug therapy within 21 days prior to enrollment
9. Unresolved toxicity from previous anticancer therapy (unless resolved to grade ≤ 1or resolved to grade 2 only if deemed clinically not significant and approved by the Sponsor) or incomplete recovery from surgery
10. Major surgery (excluding that for diagnosis) within 28 days of enrollment
11. Unstable cardiovascular function defined as:

    * Symptomatic ischemia
    * Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmic agents are excluded; first degree AV block or asymptomatic left anterior fascicular block [LAFB]/right bundle branch block [RBBB] will not be excluded), or
    * Congestive heart failure NYHA Class ≥ 3, or myocardial infarction within 3 months prior to enrollment
12. Cerebrovascular event (transient ischemic attack or stroke) within the last 12 months.
13. Major bleeding within the last 6 months.
14. Bleeding involving CNS within the last 12 months.
15. Use of any investigational agents within 30 days prior to enrollment and for the duration of the study
16. Pregnancy or lactation -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 4 months
  General safety: Vital signs (temperature, blood pressure, pulse rate, respiratory rate) and physical examination.
  • Toxicity according to the NCI CTCAE (v4.03) for AEs and clinical laboratory profile; AEs will be collected for all patients who received at least one dose of NM-IL-12 and up to one month post last NM-IL-12 dose.
Immunogenicity of NM-IL-12 | 4 months
  Immunogenicity of NM-IL-12 will be evaluated by the presence of anti-drug antibody (ADA)

SECONDARY OUTCOMES:
Response rate (Complete Response or Partial Response) as assessed by PET/CT | 4 months
  Comparison will be made between the status before salvage regimen initiation, after the second chemotherapy cycle, and after completion of all salvage chemotherapy cycles. CR and PR will be assessed according to the revised International Working Group Criteria for non-Hodgkin Lymphoma.
Time to neutrophil recovery | 4 months
  Time to neutrophil recovery, as defined by first day of ANC ≥ 500/μL
Time to platelet count recovery | 4 months
  Time to platelet count recovery, as defined by first day of self-sustained platelet count ≥ 20,000/μL
Incidence of systemic infections | 4 months
Incidence and duration of neutropenic fever | 4 months
Need for RBC and platelet transfusion | 4 months
Peak Plasma Concentration (Cmax) of NM-IL-12 | 2 months
Area under the plasma concentration versus time curve (AUC) of NM-IL-12 | 2 months
Peak Plasma Concentration (Cmax) of IFN-g and IP-10 | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yossef Kalish, MD, Principal Investigator — Hadassah Medical Organization

REFERENCES:
- [Background] Gokhale MS, Vainstein V, Tom J, Thomas S, Lawrence CE, Gluzman-Poltorak Z, Siebers N, Basile LA. Single low-dose rHuIL-12 safely triggers multilineage hematopoietic and immune-mediated effects. Exp Hematol Oncol. 2014 Apr 11;3(1):11. doi: 10.1186/2162-3619-3-11. PMID 24725395
- [Background] Gluzman-Poltorak Z, Vainstein V, Basile LA. Recombinant interleukin-12, but not granulocyte-colony stimulating factor, improves survival in lethally irradiated nonhuman primates in the absence of supportive care: evidence for the development of a frontline radiation medical countermeasure. Am J Hematol. 2014 Sep;89(9):868-73. doi: 10.1002/ajh.23770. Epub 2014 Jun 19. PMID 24852354
- [Background] Gluzman-Poltorak Z, Mendonca SR, Vainstein V, Kha H, Basile LA. Randomized comparison of single dose of recombinant human IL-12 versus placebo for restoration of hematopoiesis and improved survival in rhesus monkeys exposed to lethal radiation. J Hematol Oncol. 2014 Apr 6;7:31. doi: 10.1186/1756-8722-7-31. PMID 24708888
- [Background] Basile LA, Ellefson D, Gluzman-Poltorak Z, Junes-Gill K, Mar V, Mendonca S, Miller JD, Tom J, Trinh A, Gallaher TK. HemaMax, a recombinant human interleukin-12, is a potent mitigator of acute radiation injury in mice and non-human primates. PLoS One. 2012;7(2):e30434. doi: 10.1371/journal.pone.0030434. Epub 2012 Feb 24. PMID 22383962